CLINICAL TRIAL: NCT00518518
Title: Safety and Efficacy of Ultra-Rush High-Dose Sublingual Immunotherapy in Children With Asthma Allergic to Grass Pollen - Prospective, Randomized, Placebo Controlled Study.
Brief Title: Safety and Efficacy of Ultra-Rush Sublingual Immunotherapy in Children With Asthma Allergic to Grass Pollen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Iwona Stelmach MD, PhD, Prof, Department of Pediatrics and Allergy, Medical University of Lodz, Poland.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RNN-3-06-KE
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Asthma
Keywords: Asthma; Sublingual immunotherapy; Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Staloral 300
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Staloral 300 — Staloral 300
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The aim of the study is to assess the safety and efficacy of sublingual immunotherapy applied preseasonal and seasonal in ultra-rush scheme in children with bronchial asthma allergic to grass pollen. The investigators will assess clinical symptoms, reliever drugs usage, lung function, chosen markers of allergic inflammation, bronchial hyperreactivity with methacholine, and presence and type of allergy after two years of sublingual immunotherapy (SLIT) in children with asthma.

DETAILED DESCRIPTION:
Specific immunotherapy is the only causal treatment method of atopic diseases including bronchial asthma in children. Sublingual immunotherapy seems to be the most promising alternative to traditional specific subcutaneous injection immunotherapy.

The aim of the study is to assess the safety and efficacy of sublingual immunotherapy applied preseasonal and seasonal in ultra-rush scheme in children with bronchial asthma allergic to grass pollen. We will assess clinical symptoms, reliever drugs usage, lung function, chosen markers of allergic inflammation, bronchial hyperreactivity with methacholine, and presence and type of allergy after two years of SLIT in children with asthma.

After two years the study will be unblinded, all the children will be given grass pollen allergen extract for a year.

ELIGIBILITY:
Inclusion Criteria:

* patients allergic to grasses pollen
* patients with bronchial asthma
* patients with controlled asthma
* patients who were qualified for immunotherapy and gave written informed consent for immunotherapy

Exclusion Criteria:

* patients allergic for other perennial and seasonal allergens
* patients with other chronic diseases that either put the patient at risk when participating in the study or could influence the results of the study or the patient's ability to participate in the study as judged by the investigator

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
clinical symptoms, reliever drugs usage, controller medication usage, lung function | all visits

SECONDARY OUTCOMES:
chosen markers of inflammation (specific IgE, IgG4, eosinophils) | 1 month after baseline visit (second visit), after 5 months (fifth visit), after 18 months (ninth visit), after 30 months (thirteenth visit)
skin prick test, specific nasal provocation test with grass pollen allergen | baseline visit, after 24 months (tenth visit), after 36 months (fourteenth visit)
bronchial hyperreactivity with methacholine | after 5 months (fifth visit), after 18 months (sixth visit), after 30 months (thirteenth visit)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kaczmarek, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Poland

REFERENCES:
- [Result] Stelmach I, Kaczmarek-Wozniak J, Majak P, Olszowiec-Chlebna M, Jerzynska J. Efficacy and safety of high-doses sublingual immunotherapy in ultra-rush scheme in children allergic to grass pollen. Clin Exp Allergy. 2009 Mar;39(3):401-8. doi: 10.1111/j.1365-2222.2008.03159.x. Epub 2008 Dec 23. PMID 19134016